CLINICAL TRIAL: NCT04884347
Title: Double Blind, Randomized, Placebo-controlled Assessment of the Efficacy of a Food Supplement in Reducing Hair Loss in Male Subjects
Brief Title: Evaluation of the Efficacy of a Food Supplement in Reducing Hair Loss in Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Pharmaceutiques Trenker (Industry)
Collaborators: Complife Italia S.r.l (Unknown); Università degli Studi di Pavia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHL00.100.13.00_ IT0002110/20
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alline proMEN (Experimental): The qualitative and quantitative formula is as follows: 500 mg Keratin, 225 mg Inactive dried yeast rich in vitamin (containing 200 mg Saccharomyces cerevisiae 100% inactivated, 11.218.4 mg Vitamin B3, 6.8-7.2 mg Vitamin B5, 1.6-1.8 mg Vitamin B6, 1.6-1.8 mg Vitamin B2, 1.6 -1.8 mg Vitamin B1, 0.2-0.4 mg Vitamin B9, 0.2 mg Vitamin B8, 5.6 μg Vitamin B12), 150 mg Venus hair fern extract, 117.6 mg Iron gluconate (containing 14.7 mg Iron), 84.2 mg Sodium ascorbate coated, 76.8 mg Zinc gluconate (11 mg Zinc) 24 mg Beta carotene 20%, 14.8 mg Vitamin E, 256.3 mg Acacia gum, 100 mg Microcrystalline cellulose, 11.3 mg Magnesium stearate, 78 mg White coating (containing: 23.4-39 mg Hydroxypropylmethylcellulose (E464), 15.6-23.4 mg Calcium sulfate anhydrous (E516), 15.6-23.4 mg Magnesium carbonate, light (E504), 7.8-15.6 mg Hydroxypropylcellulose (E463), 3.9-11.7 mg Stearic acid (E570)).
  Interventions: Dietary Supplement: Alline proMEN
- Placebo (Placebo Comparator): 1095 mg Microcrystalline cellulose, 5 mg Magnesium stearate, 55 mg White coating (containing: 16.5-27.5 mg Hydroxypropylmethylcellulose (E464), 11.0-16.5 mg Calcium sulfate anhydrous (E516), 11.0-16.5 mg Magnesium carbonate, light (E504), 5.5-11.0 mg Hydroxypropylcellulose (E463), 2.8-8.2 mg Stearic acid (E570).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alline proMEN — 1 tablet per day intake during the meal with a glass of water. Treatment duration: 3 months
  Arms: Alline proMEN
Dietary Supplement: Placebo — 1 tablet per day intake during the meal with a glass of water. Treatment duration: 3 months
  Arms: Placebo

SUMMARY:
According to the American Hair Loss Association, by the age of 35, two-thirds of American men will have some degree of appreciable hair loss, and by the age of 50, approximately 50 to 85% of men will have significant hair thinning.

Hair is an essential aspect of human appearance and can have a significant impact on a person's self-esteem, mood and quality of life. Unfortunately, current treatment options can be costly, tedious or painful. They are also associated with numerous side effects.

Here, the investigators aimed at evaluating the effect of a new food supplement on hair condition in young men suffering from hair loss. A second goal was to determine tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria related to population

   * Male subjects
   * Caucasian ethnicity
   * Subjects aged between 25 and 55 years old
   * Subjects with all type of scalp and hair
   * Phototype I to IV included, according to Fitzpatrick classification
   * Subjects registered with health social security or health social insurance
   * Subjects having signed their written Informed Consent form (ICF) for their participation in the study and a photograph authorization
   * Subjects certifying the truth of the personal information declared to the Investigator
   * Subjects able to understand the language used in the investigation centre and the information given
   * Subjects able to comply with the protocol and follow protocol's constraints and specific requirements
2. Criteria related to subject's health

   * Subjects considered "healthy subject" by the Investigator
   * if the subject is under systemic pharmacological treatment, this should be stable for at least one month before the study start and do not change over the study period, excluded the treatments specified in noninclusion criteria"
3. Criteria related to hair loss disorders

   * Acute hair loss with a proportion of hair in telogen phase superior or equal to 20% as assessed by phototricogram
   * Subjects agreeing to preserve a length of hair longer than 10 cm during the study
   * Subjects agreeing to have a zone of 1.8 cm² shaved on the scalp

Exclusion Criteria:

1. Criteria related to the population

   * Subjects taking part or planning to participate to another clinical trial during the study in the same or another investigation centre
   * Subjects deprived of freedom by administrative or legal decision or under guardianship Subjects not able to be contacted in case of emergency.
   * Subjects admitted in a sanitary or social facility
   * Subjects planning a hospitalisation during the study
   * Subjects belonging to the staff of the investigation centre
   * subjects who have participated in another clinical trial with anti-hair loss product or treatment within the last 12 weeks before the inclusion visit
2. Criteria related to subject's health

   * Subjects having an acute, chronic or progressive illness liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
   * Subjects being in course of a long-treatment or intending to have one, in particular with aspirin, products containing aspirin, corticoids, beta blockers (including eye drops), immuno-suppressive and/or desensitisation drugs or under any treatment considered by the Investigator liable to interfere with the study data or incompatible with the study requirements
   * Subjects being vaccinated within the 3 weeks prior to the study or intending to be vaccinated during the course of the study
   * Subjects having a skin condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements Subjects having personal history of cosmetic, drug or domestic products irritative reactions Subjects having personal history of cosmetic products or adhesive plaster allergy Subjects having personal history of drug, domestic products and food allergy with no progressive or recent clinical features of allergy
3. Criteria related to hair loss disorders

   * Subjects who have any other diagnosed hair disorder or hair disease.
   * Subjects having excessive and/or fluctuating hair shedding for more than 6 months Subjects with Inflammatory skin disease or progressive skin lesion on the scalp (psoriasis, seborrhoeic dermatitis, severe erythema, severe excoriation, severe sunburn, etc.). Subjects having a scalp lesion in relief which may be traumatized
   * Subjects with history of hypersensitivity or intolerance to any of the following components applied by topical route: ethyl alcohol, components of the used hair dye, components of the studied product.
   * Subjects having systemic treatment affecting the hair growth taken for more than 4 consecutive weeks during the last 24 weeks before inclusion visit: Retinoids, Anti-mitotic, cytotoxic drugs other than antineoplastic, Anti-androgens (spironolactone, flutamide), androgens, Anti-epileptic agents, interferon alpha
   * Subjects having systemic or local androgenetic alopecia treatment or product, taken or applied (Minoxidil, Aminexil, Finasteride, Dutasteride, cosmetic solution or capsules with vitamin B, zinc, caffeine…) for more than 4 consecutive weeks during the last 24 weeks before the inclusion visit
   * Subjects having any other local treatment applied on the scalp (non-steroidal anti-inflammatory, ketoconazole…) within the last 2 weeks before the inclusion visit
   * Subjects having any following hair care within the last 2 weeks before the inclusion visit or foreseen during the study (except for dying): dandruff shampoo, antifungal shampoo, dyeing, bleaching, perm
   * Subjects having any hair care product applied on the scalp between the last shampoo and the inclusion visit (e.g. gel, hairspray, wax, foam…)
   * Subjects under radiotherapy, chemotherapy at any time Subjects having scalp surgery (hair transplants, laser) at any time

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the number of hair in anagen and telogen phases at day 30 and 86. | Day 0, Day 30, Day 86
  The total number of hair (hair density) and the number of hair in the anagen phase will be determined by phototricogram. Briefly, all hairs in a 2 sq cm area are trimmed 1 mm from the skin surface. The hair is dyed and a baseline photograph is taken. After 48h, the same region is photographed again. By comparing with the baseline picture, one can observe as to which hair fibers have grown (follicles in anagen) and which have not (follicles in telogen) and the density of the hair (the number of hairs in the photograph). Anagen hair will be manually counted comparing side by side the photographs taken at each checkpoint and 48 hours after. Telogen hair will be calculated as the difference between the total hair number and the anagen hair number.

SECONDARY OUTCOMES:
Changes from baseline in hair radiance (au) at day 28 and day 84 | Day 0, Day 28, Day 84
  Hair radiance will be measured by spectrophotometry.
Changes from baseline in hair elongation (%) at day 28 and day 84 | Day 0, Day 28, Day 84
  Hair elongation (hair elasticity) will be evaluated by means of dynamometer reading. The dynamometer reading will be done on a single hair fiber. In total 10 hair fibers/participant will be measured.
Changes from baseline in hair breakage force (cN) at day 28 and day 84 | Day 0, Day 28, Day 84
  The force at which the hair breaks (breakage force) will be evaluated by means of dynamometer reading. The dynamometer reading will be done on a single hair fiber. In total 10 hair fibers will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Nobile, PhD, Study Director — Complife Italia S.r.l
Locations (1):
- Complife Italia S.r.l, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No